CLINICAL TRIAL: NCT03949205
Title: Effects of Breaks of Sedentary Behavior With Isometric Exercise in Cardiovascular Health Indicators of Adults
Brief Title: Sedentary Behavior Breaks With Isometric Exercise in Cardiovascular Health Indicators
Acronym: BREAK001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Raphael Mendes Ritti Dias, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BREAK001
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Sedentary Behavior
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial and randomized crossover trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leg Extension Isometric Training (Experimental): Experimental group will perform leg extension isometric exercise.
  Interventions: Other: Leg Extension Isometric Training
- Control Group (No Intervention): Control group will be advised to maintain their work habits and not to change their routine activities, especially diet and physical activities.

INTERVENTIONS:
Other: Leg Extension Isometric Training — The leg extension isometric exercise will be performed tree times a week , in four 2 min bouts of isometric contraction, at a intensity of 30% of maximal voluntary contraction and an interval of two minutes between bouts.
  Arms: Leg Extension Isometric Training

SUMMARY:
The goal of this study is to analyze the chronic effects of sedentary behavior breaks using the leg extension isometric exercise in the cardiovascular health indicators of healthy adults exposed to prolonged time in the sitting position. The patients recruited will be randomized into two groups: leg extension isometric training (TIE) and control group (CG). The TIE group will perform 12 weeks of isometric training. The CG will be advised not to change their routine activities, especially diet and physical activities.In the pre and post-intervention periods cardiovascular measures will be obtained.

DETAILED DESCRIPTION:
Long periods in sedentary behavior promote deterioration of vascular function, which is directly associated with the occurence of chronic noncommunicable diseases. In this context, the execution of interruptions in this behavior (breaks) is recommended. Studies have shown benefits of isometric training in vascular function, which could be useful to minimize the consequences of time spent in sedentary behavior. Thus, the goal of this study is to analyze the chronic effects of sedentary behavior breaks using leg extension isometric exercise in the cardiovascular health indicators of adults exposed to prolonged time in the sitting position. The target population of the study will consist of healthy subjects above 18 years of age of both genders. All subjects will be submitted to measurements of endothelial function, blood pressure and cardiac autonomic modulation. After these measurements, the subjects will be randomized into two groups: leg extension isometric training group (TIE) and control group (CG). After 12 weeks both groups will be submitted to the same measurements from pre-intervention.

ELIGIBILITY:
Inclusion Criteria:

* No diagnostic of cardiovascular diseases or diabetes
* Do not present high cardiovascular risk
* Do not participate in an exercise program in the previous six months
* Occupational activity that requires more than six hours of sitting time per day
* Do not be a smoker or make use of medications

Exclusion Criteria:

* Adherence to the training sessions inferior to 85%
* Adherence to another supervised exercise program
* Change the characteristics of the occupational activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in vascular function at 12 weeks | Baseline and 12 weeks
  Vascular function will be measured before and after 12 weeks of intervention on the intervention and control groups by a bidimensional ultrasonography device with spectral Doppler and linear transducer.

SECONDARY OUTCOMES:
Changes from baseline in blood pressure at 12 weeks | Baseline and 12 weeks
  Blood pressure will be measured before and after 12 weeks of intervention period on intervention and control group by an automatic blood pressure monitor (HEM-742, Omron Healthcare, Japan).
Change from baseline in cardiac autonomic modulation at 12 weeks | Baseline and 12 weeks
  Cardiac autonomic modulation will be measured before and after 12 weeks of intervention period on intervention and control group by heart rate monitor (Polar V800, Polar Electro, Finland).

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Ritti-Dias, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the data upon requirement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 1 year after the end of recruitment.